CLINICAL TRIAL: NCT00435435
Title: Phase Four Randomized, Multicentre, Open-Label, Comparative Trial Of Disulfiram, Nalterexone And Acamprosate In The Treatment Of Alcohol Dependence
Brief Title: Comparative Trial Of Disulfiram, Naltrexone And Acamprosate In The Treatment Of Alcohol Dependence
Acronym: DNA
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Finnish Institute for Health and Welfare (Other Government)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KTL-175-1
Record Dates: First submitted 2007-02-14; First posted 2007-02-15 (Estimated); Last update posted 2007-02-16 (Estimated); Status verified 2000-02

CONDITIONS: Alcohol Dependence
Keywords: Alcoholism; Dependence; Randomization; Effect; Disulfiram; Naltrexone; Acamprosate
MeSH Terms: conditions — Alcoholism | interventions — Disulfiram; Acamprosate

INTERVENTIONS:
Drug: Disulfiram
Drug: Acamprosate
Drug: Naltexone

SUMMARY:
The aim of this study was to compare the effect of manual based cognitive therapy in adjunct of three different pharmacotherapy.

DETAILED DESCRIPTION:
Context Alcoholism is common clinical problem and its treatment has no standard and is controversy. Different pharmacotherapy's, acamporsate, nalterxone and disulfiram have shown to improve the drinking outcomes, but there is no randomized comparative studies on the effects of these three medications.

Objectives The aim of this study was to compare the effect of manual based cognitive therapy in adjunct of three different pharmacotherapy.

Design and setting Randomized, open label, multicentre naturalistic study, 12 week continuous medication followed by targeted medication up to 52weeks and 67 week follow up on voluntary treatment seeking alcohol dependent outpatients.

Participants 243 alcohol dependent adults. Intervention Subjects were randomized 1:1:1 to receive naltrexone, acamprosate or disulfiram, 50 mg, 1998 mg or 200 mg correspondingly per day. The patients were met weekly in first month, then after 3, 6 and 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Alcohol dependence (ICD-10)

Exclusion Criteria:

* Clinically significant symptoms of alcohol withdrawal
* Significant recently diagnosed psychiatric disease (psychosis, personality disorder or suicidal tendency that appeared during the initial interview)
* Current psychiatric disease demanding special treatment or medication including DSM-IV determined drug dependence other than alcohol or nicotine dependence
* Current use of any opioids within four weeks before screening
* Significant brain, thyroid, kidney, uncompensated heart disease, or clinically significant liver disease (cirrhosis, aqlcoholic hepatitis or ALAT > 200)
* Pregnancy, nursing, or women refused to use a reliable method for birth control

Ages: 25 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 243
Dates: Start 2000-09; Study Completion 2005-04

PRIMARY OUTCOMES:
Time(days) to first heavy drinking (HDD)day after medication started

SECONDARY OUTCOMES:
Time (days) to first drinking after medication started
Abstinence days (0 drinks/ day) by group
Average alcohol intake (weekly by group)
ALAT
GGT
SADD
AUDIT
EQ-5

CONTACTS AND LOCATIONS:
Overall Officials: Hannu Alho, MD, PhD, Study Director — National Public Health Institute, Department of Mental health and Alcohol Research
Locations (1):
- National Public Health Institute, Department of Mental Health and Alcohol Research, Helsinki, Finland

REFERENCES:
- [Background] Morley KC, Teesson M, Reid SC, Sannibale C, Thomson C, Phung N, Weltman M, Bell JR, Richardson K, Haber PS. Naltrexone versus acamprosate in the treatment of alcohol dependence: A multi-centre, randomized, double-blind, placebo-controlled trial. Addiction. 2006 Oct;101(10):1451-62. doi: 10.1111/j.1360-0443.2006.01555.x. PMID 16968347